CLINICAL TRIAL: NCT05504876
Title: A Single-center, Open-label Study to Investigate the Effect of a Single Oral Dose of HEC74647 and HEC110114 on the Pharmacokinetics of Midazolam, and Their Metabolites in Healthy Subjects
Brief Title: Pharmacokinetics of Midazolam When Co-administered With HEC74647 and HEC110114
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEC74647/HEC110114-DDI-101
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Midazolam Syrup HEC74647PA HEC110114 (Experimental): Subjects will receive 5mg Midazolam Syrup on Day 1,100 mg HEC74647PA and 600 mg HEC110114 on Day3~8, 5mg Midazolam Syrup co-administered with 100 mg HEC74647PA and 600 mg HEC110114 on Day9.
  Interventions: Drug: Midazolam Syrup; Drug: HEC74647PA; Drug: HEC110114

INTERVENTIONS:
Drug: Midazolam Syrup — Administered Midazolam Syrup 5 mg orally once daily in fed state;
Drug: HEC74647PA — Administered HEC74647PA 100 mg orally once daily in fed state;
Drug: HEC110114 — Administered HEC110114 600 mg orally once daily in fed state;

SUMMARY:
This is a single center, open-label study to investigate whether HEC74647 and HEC110114 has an effect on the pharmacokinetic (PK) profile of midazolam（a cytochrome (CYP) 3A4 substrate）in healthy subjects

DETAILED DESCRIPTION:
This is a single center, open-label study in healthy adult subjects. Total 14 subjects will be enrolled into the study and will be receive study drug per the defined treatment.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form before the trial and fully understand the contents of the trial, the process and possible adverse reactions.
* Be able to complete the study according to the trail protocol.
* Subjects (including partners) have no pregnancy plan within 3 months after the last dose of study drug and voluntarily take effective contraceptive measures.
* Must be male or female between 18 to 45 years of age inclusive.
* Male and female should weigh no less than 50 kg and 45 kg respectively, and body mass index (BMI) between 18 and 28 kg /m2, inclusive.
* Physical examination and vital signs without clinically significant abnormalities.

Exclusion Criteria:

* Use of >5 cigarettes per day during the past 3 months.
* Known history of allergy to study drugs#or allergies constitution ( multiple drug and food allergies
* History of alcohol abuse (14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits or 100 mL of wine).
* Donation or loss of blood over 450 mL within 3 months prior to screening.
* 12-lead ECG with clinically significant.
* Positive for Viral hepatitis (including hepatitis B and C), HIV and syphilis.
* Subjects deemed unsuitable by the investigator for any other reason.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Effect of Steady-state Oral HEC74647PA and HEC110114 on the Single Dose Pharmacokinetics (PK) of Oral Midazolam in Healthy Subjects (Cmax) | Day 1, Day9
Effect of Steady-state Oral HEC74647PA and HEC110114 on the Single Dose Pharmacokinetics (PK) of Oral Midazolam in Healthy Subjects (AUC0-t) | Day 1, Day9
Effect of Steady-state Oral HEC74647PA and HEC110114 on the Single Dose Pharmacokinetics (PK) of Oral Midazolam in Healthy Subjects (AUC0- 0-∞) | Day 1, Day9
Incidence of adverse eventsECG, or Physical Examination. | Day 1 to Day16

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Hong, Doctor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China